CLINICAL TRIAL: NCT01428492
Title: A Phase Ib Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the Oral AKT Inhibitor GSK2110183 Administered in Combination With Bortezomib and Dexamethasone in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Ph 1b Study to Evaluate GSK2110183 in Combination With Bortezomib and Dexamethasone in Subjects With Multiple Myeloma
Acronym: PKB115125
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115125
Record Dates: First submitted 2011-08-11; First posted 2011-09-05 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: AKT Inhibitor; hematologic malignancies; GSK2110183; bortezomib; multiple myeloma; dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — GSK2110183; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1-Dose Escalation (Experimental): GSK2110183 is administered in combination with bortezomib and dexamethasone until MTD is met.
  Interventions: Drug: GSK2110183; Drug: Bortezomib; Drug: Dexamethasone
- Part 2- Pharmacokinetic/Pharmacodynamics Cohort (Experimental): Once the MTD(s) has been determined, up to 9 subjects of the total enrolled in Part 2 will be entered in the Pharmacokinetic/Pharmacodynamic Cohort. Subjects will be enrolled in this cohort to explore whether exposure to GSK2110183 at dose identified in Part 1 is similar when GSK2110183 is administered alone or in combination with bortezomib and dexamethasone. The same relationship will be explored for bortezomib and dexamethasone when the two drugs are give alone or in combination with GSK2110183.
  Interventions: Drug: GSK2110183; Drug: Bortezomib; Drug: Dexamethasone
- Part 2- Safety/Clinical Activity Cohort (Experimental): Enrolment into the safety/clinical activity cohort in Part 2 will begin prior to enrollment in the PK/PD cohort. Subjects with relapsed multiple myeloma who are either bortezomib sensitive or naive after failing one line of prior systemic therapy will be enrolled in the Safety/Clinical Activity cohort. "Bortezomib sensitive" is defined as having a response (PR or better) to the last bortezomib-containing therapy lasting at least 60 days beyond the end of therapy. A minimum of 15 subjects and a total of 40 subjects will be enrolled. This expansion cohort will further characterize the safety and clinical activity profile of GSK2110183 to inform the future development of this combination regimen.
  Interventions: Drug: GSK2110183; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: GSK2110183 — The oral, once daily dose of GSK2110183 will be dependent on the cohort to which a subject is assigned. Subjects enrolled in Cohort 1 will receive 75 mg GSK2110183 once daily. Dose escalation in Schedule A and Schedule B will follow 25 mg increments in a 3+3 dose escalation procedure up to a maximum of 150mg daily or until MTD is reached, whichever comes first, for each schedule. GSK2110183 will continue at daily dosing until treatment discontinuation criteria is met.
Drug: Bortezomib — Bortezomib (1.0 mg/m2) will be administered on days 1, 4, 8, and 11 of each 21-day cycle for cohort 1 for up to 8 cycles. Bortezomib (1.3 mg/m2) will be administered on days 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles. Bortezomib (1.5 mg/m2) will be administered on days 1, 8, and 15 of each 21-day cycle for up to 8 cycles.
Drug: Dexamethasone — Dexamethasone will be given orally at a fixed dose of 20 mg only on days of bortezomib dosing in both Schedule A and Schedule B.

SUMMARY:
Phase Ib, open-label study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and clinical activity of GSK2110183 dosed in combination with bortezomib and dexamethasone in multiple myeloma (MM) subjects who have failed at least one line of systemic treatment. Part 1 will identify the maximum tolerated dose(s) (MTD) of the combination regimen. Schedule A - GSK2110183 administered once daily with bortezomib (1.3 mg/m2) and dexamethasone (20 mg) given biweekly. Part 2 will further explore the safety, tolerability and clinical activity of the MTD(s) identified in Part 1, including a pharmacokinetic cohort.

DETAILED DESCRIPTION:
This is a Phase Ib, open-label study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and clinical activity of GSK2110183 dosed in combination with bortezomib and dexamethasone in relapsed/refractory multiple myeloma (MM) subjects who have failed at least one line of systemic treatment. Part 1 will identify the maximum tolerated dose(s) (MTD) of the combination regimen.

Part 1, Schedule A will assess the safety and pharmacodynamics of GSK2110183 administered once daily with bortezomib (1.3 mg/m2) and dexamethasone (20 mg) given biweekly. It is estimated that up to 35-45 evaluable subjects will be enrolled in Part 1. Part 2 will explore further the safety, tolerability, pharmacokinetics, pharmacodynamics and clinical activity of the MTD(s) identified in Part 1. A minimum of 15 and maximum of 40 subjects will enroll in Part 2 Safety/Clinical Activity Cohort for each Schedule explored. The Part 2 PK/PD cohort will enroll up to 18 subjects. This pharmacokinetic cohort will explore whether exposure to GSK2110183 at the MTD is similar when GSK2110183 is administered alone or in combination with bortezomib and dexamethasone. The same relationship will be explored for bortezomib and dexamethasone when the two drugs are given by themselves or in combination with GSK2110183. The identified MTD(s) and pharmacodynamic results in this study will inform the doses for future development of the regimen of GSK2110183 dosed in combination with bortezomib and dexamethasone in subjects with relapsed/refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 18 years or older.
* Performance status score of 0 - 2 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain oral medication.
* Histologically confirmed diagnosis of Multiple Myeloma (MM). Subjects enrolled in the Safety/Clinical Activity Cohort (Part 2) must have relapsed MM (bortezomib-naive or bortezomib sensitive) with at least one of the following: Serum M-protein ≥1.0g/dl (≥10gm/l); Urine M-protein ≥200 mg/24h; Serum Free Light Chain (FLC) assay: Involved FLC level ≥5mg/dl (≥50mg/l) and an abnormal serum free light chain ratio (<0.26 or >1.65); Biopsy proven plasmacytoma (should be measured within 28 days of Screening Visit)
* Failed at least 1 line of systemic therapy. The preparative regimen (with or without total body irradiation) and subsequent autologous stem cell rescue used for an autologous stem cell transplant are considered as one line of therapy.
* Subjects with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met:
* transplant was > 100 days prior to study enrolment
* no active infection
* subject meets the remainder of the eligibility criteria outlined in this protocol
* Fasting serum glucose <126 mg/dL (<7 mmol/L). Subjects diagnosed previously with Type 2 diabetes must also meet the additional following criteria:
* Diagnosis of diabetes ≥6 months prior to enrolment
* HbA1c≤8% at Screening visit
* Adequate organ system function as defined in protocol.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e. physiologically incapable of becoming pregnant) defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MIU/ml and estradiol <40 MIU/ml and estradiol <40 pg/ml (<147pmol/L) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential, has a negative serum pregnancy test during the screening period, and agrees to use one of the contraception methods in protocol from screening until four weeks after the last dose of study drug.
* Male subjects with female partners of childbearing potential must have had a prior vasectomy or agree to use one of the contraception methods in protocol. This must be followed from the time of the first dose of study drug until 3 months after the last dose of study drug.

Exclusion Criteria:

* Chemotherapy, radiotherapy, immunotherapy, or other anti-myeloma therapy within 14 days prior to the first dose of any one of the drugs in the combination regimen. In addition, any drug-related toxicity should have recovered to Grade 1 or less.
* Use of an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of any one of the drugs in the combination regimen.
* History of an allogeneic stem cell transplant. Subjects with a history of an autologous stem cell transplant are NOT excluded if they meet Inclusion Criteria #7.
* Current use of prohibited medication listed in the protocol during treatment with GSK2110183.
* Current use of oral corticosteroids, with the exception of inhaled or topical steroids. Dexamethasone will be given only in combination with bortezomib on this study.
* Anticoagulants are permitted only if the subject meets Partial Thromboplastin Time (PTT) and International Normalized Ratio (INR) entry criteria. Their use must be monitored in accordance with local institutional practice.
* Presence of active gastrointestinal disease or other condition that could affect gastrointestinal absorption (e.g. malabsorption syndrome) or predispose subject to gastrointestinal ulceration.
* Evidence of mucosal or internal bleeding.
* Presence of > Grade 1 peripheral neuropathy at screening.
* Unresolved toxicity (except alopecia) ≥ Grade 2 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 [NCI-CTCAE, 2009] from previous anti-cancer therapy.
* Any major surgery within the last four weeks.
* Type 1 diabetes mellitus.
* Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject's safety or providing informed consent.
* Known active infection requiring parenteral or oral anti-infective treatment.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease, unstable hypertension).
* Primary or metastatic malignancy of the central nervous system.
* Previous or concurrent malignancies are allowed if it is clear that the other tumor is not contributing to the subject's illness. The subject must not be receiving active therapy for this disease and the disease must be considered medically stable..
* QTc interval ≥ 470 msec
* Other clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening.
* Class III or IV heart failure as defined by the New York Heart Association (NYHA) (1994) functional classification system.
* Known hypersensitivity to any of the components of the study treatment.
* Pregnant or lactating female.
* History of known HIV infection.
* Subjects with a positive test for Hepatitis C (HCV) antibody are excluded, regardless of viral load. If hepatitis C antibody is positive, confirmatory tests may be performed.
* History of "active" Hepatitis B (HBV) infection. Hepatitis B carriers are eligible only if antiviral therapy is administered as outlined in the guidelines in the protocol. Hepatitis B carrier is defined as HBsAg and HBcAb positive by liver enzymes (AST and ALT) are normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The recommended Phase II dose (RP2D) and schedule of GSK2110183, bortezomib and dexamethasone dosed in combination. | Estimation is that each subject may be assessed for up to 48 months.
  Dose and schedule determined using adverse events and changes in safety assessments (laboratory parameters, vital signs and ECG parameters). Recommended Phase 2 Dose (RP2D) will be defined in Part 1. The specific number of subjects to be enrolled is dependent on the number of dose limiting toxicities (DLTs) reported; enrollment of up to 45 subjects in Part 1 is estimated. Subjects will continue on study from the date of randomization until the date of the first documented disease progression or when the subject meets one of the Treatment Discontinuation criteria, whichever comes first

SECONDARY OUTCOMES:
Pharmacokinetics of GSK2110183, bortezomib and dexamethasone. Composite (or Profile) of Pharmacokinetics Time Frame: predose, 0, 5 min, 15 min, 1, 2, 3, 4, 6, 8, 10-12, 14-22, and 24 hrs post-dose. | Part 2, PK plasma samples will be collected on Cycle 0 Day 11 and Day 38 and Cycle 1 Day 11 (each day at predose, 5min, 15min, 1, 2, 3, 4, 6, 8, 10-12, 14-22 and 24 hrs). Part 1 and Part 2, 3 PK plasma samples will be collected on Day 1 of Cycles 2 - 8
  Comparison of GSK2110183 area under the concentration versus time curve (AUC) values when administered alone versus when administered with bortezomib and dexamethasone. Comparison of bortezomib and dexamethasone AUC values when administered alone versus when administered with GSK2110183. Comparison of GSK2110183 maximum concentration (Cmax) values when administered alone versus when administered with bortezomib and dexamethasone. Comparison of bortezomib and dexamethasone Cmax values when administered alone versus when administered with GSK2110183.
Clinical activity | Lab assessment of disease (i.e., quantitative paraprotein, SPEP/UPEP) occurs at beginning of cycles, or every 3 wks. Extramedullary disease assessed every 12 wks by imaging, only as warranted.
  The clinical response [ i.e. changes in the M-protein, the serum free light chains (FLC) (kappa/lambda ratio ), the appearance of or the change in the size of plasmacytomas or lytic lesions in bone ] to GSK2110183, bortezomib and dexamethasone in subjects with relapsed/refractory multiple myeloma, as assessed by the International Myeloma Working Group Uniform Response Criteria
Relationships between GSK2110183, Pharmacokinetic (PK), Pharmacodynamic (PD) and clinical activity. Composite (or Profile) of Serial Pharmacokinetics Time Frame: predose, 5 min, 15 min, 1,2,3,4,6,8, 10-12, 14-22, and 24 hours post-dose. | Part 2, serial PK plasma samples will be collected on Cycle 0 Day 11 and Day 38 and Cycle 1 Day 11. In Part 1 and 2, PD markers (BM biopsy and aspirite, plasma for cfDNA and CAF) will be collected predose, once post dose and at time of relapse.
  Explore the relationships between GSK2110183 exposure (AUC, Cmax concentration, minimum concentration), PD markers (e.g., changes in phosphorylation of markers of AKT (pAKT) pathway activation in bone marrow (BM) biopsy samples and clinical activity (M Protein levels, clinical response). In Part 2, Serial PK plasma samples collected on 2 days. Parts 1 and 2, samples for PD markers (BM biopsy and/or aspirate, plasma for circulating free DNA (cfDNA) or cytokine and angiogenic factors (CAFs)) collected. Parts 1 and 2, clinical activity (lab assessments, quantitative paraprotein) assessed.
Exploratory Translational Research | BM biopsy for AKT activation markers (predose, once post dose). Plasma for cfDNA and CAFs (predose, once post dose, at time of relapse). BM aspirate to assess potential predictive markers of response: FISH (predose) and cytogenetics (predose and CR).
  Phosphorylation of markers of AKT pathway activation (i.e., pAKT and pPRAS40) in bone marrow biopsy samples. Exploratory analysis of potential predictive markers of response [i.e., cytogenetics (CD45, CD138, CD38, CD19, CD56, CD20, CD117), FISH [t(4;14), t(14;16), 17p13del, del(13q)], Ki67, mutations in NRAS and KRAS] and soluble cytokine levels (i.e., VEGF, IL-6, IFG1) in plasma. BM biopsy will assess markers of AKT activation. Plasma samples will assess circulating free DNA and CAFs. BM aspirate will assess potential predictive markers of response collected for FISH and cytogenetics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (8):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
- Novartis Investigative Site, Galway, Ireland
- Novartis Investigative Site, Taipei, Taiwan